CLINICAL TRIAL: NCT03717285
Title: Under Direct Vision Versus Under Non Direct Vision for The Efficacy and Safety Ureteral Access Sheath in RIRS for the Management of ≤20mm Size Kidney Stones: A Single-center Randomized Controlled Trial
Brief Title: Under Direct Vision vs Under Non Direct Vision of Insertion of UAS in RIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MRER(75)2018
Record Dates: First submitted 2018-10-07; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Urolithiasis
Keywords: RIRS; Renal stones; ureteral access sheath; ureteral injury
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:Under direct vision (Experimental): Patients in Group 1 insert the UAS under direct vision.In this procedure,the investigators will insert the ureteroscope into urinary bladder beside the guidewire to observe the process of uas insertion into the ureter.
  Interventions: Procedure: Insert the UAS under direct vision
- Group 2:Under non direct vision (Active Comparator): Patients in Group 2 insert the UAS under non direct vision.In this procedure,the investigators will insert the UAS under fluoroscopy control.
  Interventions: Procedure: Insert the UAS under non direct vision

INTERVENTIONS:
Procedure: Insert the UAS under direct vision — Patients in this group，we use rigid ureteroscopy to insert the UAS under direct vision.
  Arms: Group 1:Under direct vision
Procedure: Insert the UAS under non direct vision — Patients in this group，we insert the UAS by the experience of the surgeon and under non direct vision .
  Arms: Group 2:Under non direct vision

SUMMARY:
Retrograde intrarenal surgery (RIRS) has been considered as the first-line choice for the management of <20mm kidney stones. Insertion of a ureteral access sheath (UAS) before RIRS surgery is currently accepted as an effective method to improve the effectiveness of surgery, but can be accompanied by serious complications. In long-term clinical practice， the investigators has found that many ureteral injuries occur during UAS insertion of the ureter from ureteral orifice. And if we use rigid ureteroscopy to insert the UAS under direct vision, we can provide the placement success rate and reduce the incidence of complications. The investigator aims to perform a prospective and randomized controlled trial comparing the safety and efficacy of under direct vision and under non direct vision during the insertion of UAS.

DETAILED DESCRIPTION:
Retrograde intrarenal surgery (RIRS) has been considered as the first-line choice for the management of <20mm kidney stones. Insertion of a ureteral access sheath (UAS) before RIRS surgery is currently accepted as an effective method to improve the effectiveness of surgery, but can be accompanied by serious complications. In long-term clinical practice， the investigators has found that many ureteral injuries occur during UAS insertion of the ureter from ureteral orifice. And if we use rigid ureteroscopy to insert the UAS under direct vision, we can provide the UAS insertion success rate and reduce the incidence of complications.

Options for the UAS insertion include inserted under fluoroscopy control or inserted by the experience of the surgeon. The former is more commonly used in the United States, while the latter is more commonly used in China. But neither is perfect. Moreover, Ibrahim Karabulut et al. and Mehmet Giray Sönmez et al. reported a different technique for placement ureteral access sheath called "Endovisional technique" in which the outer sheath of UAS was worn on the semirigid endoscope and placed into the ureter under direct vision. Nevertheless, They found that complication rate was lower in the patients who had the UAS placed under "Endovisional technique" when compared to the classical technique. But the difference was not statistically significant. In addition, the investigators are concerned that failure to use sheath cores may cause new damage to the ureter.

So the investigators find a new way to insert UAS without damaging the ureter. In our new procedure, the patient is placed in the lithotomy position, and a 0.035'' flexible tip guidewire is placed into the renal pelvis using a ureteroscope. Then take out the ureteroscope and insert the ureteroscope into urinary bladder beside the guidewire. A 12 Fr/ 14 Fr ureteral access sheath (UAS) is advanced into the ureteral over the guidewire under direct vision. When the UAS successfully enters the ureteral orifice a few centimeters, the ureteroscope is removed. Continue inserting the UAS into the proximal ureter or UPJ and use the direct urinary system X-graphy (DUSG) to confirm that the UAS is inserted into the correct position. A P5 or P6 Olympus flexible ureteroscope is passed through the UAS to finish lithotripsy.

Until now, routine technique to insert ureteral access sheath during RIRS is still under discussion. The investigator aims to perform a prospective and randomized controlled trial comparing the safety and efficacy of under direct vision and under non direct vision during the insertion of UAS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be a suitable operative candidate for RIRS
2. Age 18 to 70 years
3. Normal renal function 4 .ASA score Ⅰ and Ⅱ

5. Single renal stone ≤20mm or multiple stones the conglomerate diameter (additive maximal diameter of all stones on axial imaging of computed tomography) up to 20 mm

Exclusion Criteria:

1. Patients with solitary kidney
2. Uncorrected coagulopathy and active urinary tract infection (UTI)
3. Prior ipsilateral endourological procedure history, such as RIRS, PCNL, URS and URL
4. Patients who underwent transplant or urinary diversion.
5. Congenital abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-09-10 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
UAS insertion success rate | intraoperatively
  Primary insertion of a UAS is not always possible. The ideal position of the UAS is with its distal extremity just below the ureteric-pelvic junction (UPJ). Insertion failure is defined as UAS cross the upj or do not reach the proximal ureter or the surgeon's decision to resign UAS insertion due to high resistance to the retrograde progression of the UAS along the urinary tract.

SECONDARY OUTCOMES:
Complication rate | 1 month after removing the pigtail stent
  Complication is defined as any adverse event occurred intraoperatively or ≤1 month postoperatively, including intraoperative bleeding, postoperative pain and so on.The investigator will invaluate perioperative complications by modified Clavien system
Ureteral lesion grade | intraoperatively
  Base on post-ureteroscopic lesion scale (PULS), reported byTraxer O and Thomas A in 2013.UAS related ureteral injuries were divided into 5 grades according to ureteral wall anatomy.Grade 0 means no lesion found or only mucosal petechiae. Grade 1 means ureteral mucosal erosion without smooth muscle injury. Both Grade 0 and Grade 1 are considered as low-level injuries. Grade 2 means ureteral wall injury, including mucosa and smooth muscle, with adventitial preservation (periureteral fat not seen). Grade 3 means ureteral injury indicated ureteral perforation involving the full thickness of the ureteral wall, including the adventitia.Grade 4 means injury corresponded to total ureteral avulsion with complete rupture of ureteral continuity. Grade 2, 3 and 4 are high-level injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, Ph.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- epartment of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China